CLINICAL TRIAL: NCT02733003
Title: Implementation Research for Vulnerable Women in South Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: Kheth'Impilo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: R01AA022882 (NIH)
Record Dates: First submitted 2016-01-21; First posted 2016-04-11 (Estimated); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: HIV; Substance Abuse
Keywords: Implementation Science; HIV; Sexual Risk; Sexually Transmitted Diseases; Substance Abuse; Violence and Victimization; Linkage to care; Gender-based Violence; Antiretroviral Therapy (ART)
MeSH Terms: conditions — Substance-Related Disorders; Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Women's Health CoOp (WHC) (Experimental): This is an adapted behavioral intervention for women in South Africa, who use alcohol and other drugs and are living with HIV or at risk of acquiring HIV.
  Interventions: Behavioral: Women's Health CoOp (WHC)

INTERVENTIONS:
Behavioral: Women's Health CoOp (WHC) — Participants in this group will participate in two workshops of the woman-focused intervention about HIV/STIs, sexual behaviors, alcohol and other drug use, violence, communication skills, and other issues.

SUMMARY:
This study sought to implement the Women's Health CoOp (Cooperative) (WHC) intervention into healthcare, antenatal, and substance treatment clinics in South Africa and translated this evidence-based intervention into real-world settings. Implementation, service, and patient outcomes will be evaluated through an iterative stepped wedge design.

DETAILED DESCRIPTION:
This five-year implementation science study used a cluster-randomized stepped-wedge design to evaluate the implementation, service, and patient outcomes associated with the WHC for alcohol and other drug (AOD)-using HIV positive women in usual care settings.

A list of four substance use treatment clinics and four healthcare clinics, identified and approved by the City of Cape Town, South Africa were randomized to begin the intervention during one of the four cycles. Each healthcare clinic was paired with a substance use treatment clinic based on geographic proximity, and each pair was randomized by computer into four succeeding 6-month implementation cycles where implementation of the WHC took place simultaneously at the paired sites. Approximately 120 HIV positive participants were recruited in each cycle (approximately 60 from each clinic) for the patient level outcomes.

Both qualitative and quantitative data were collected to assess the appropriateness of marketing plans developed through formative methods, as well as the acceptability, adoption, feasibility, fidelity, and sustainability of the WHC intervention implementation as well as service outcomes (comprehensive services and timely service linkages) during each implementation cycle.

Each implementation cycle included a pre-implementation period, implementation period (6-months), and post-implementation period. In the pre-implementation period, focus groups and questionnaires surveys were conducted with clinic staff to assess the readiness of each site to implement the WHC. During the implementation period, employees at each site were trained to facilitate the WHC and the WHC was integrated into site operations. Subsequently, in the post-implementation period the researchers collected data related to challenges, benefits, and sustainability from each site. The process was repeated for each cycle and these formative periods between cycles were used to inform backward- and forward- implementation strategies, make modifications to the WHC, and leave time for site-specific training for the next cycle. Consequently, the sites randomized to the first cycle had the longest post-intervention observation period whose implementation sustainability was checked through fidelity forms and sustainability questionnaires, and sites in the fourth cycle benefited the most because of lessons learned and information shared from previous cycles.

The intervention was implemented in a group, however there were instances when only one participant was available and therefore the intervention was implemented one-on-one. The WHC has previously been tested in group and one-on-one formats and both have demonstrated consistent significant intervention effects. Research staff trained clinic staff members to deliver the intervention. The intervention was delivered by clinic staff and was not part of the research. The research questions were related to the feasibility of implementing the intervention in clinics and its acceptability to clinic staff and patients. The researchers collected information on patient-level outcomes to determine if the intervention was effective when it was delivered by clinic staff to patients in the clinic. Also, to assess acceptability of the intervention workshops among patients, the researchers conducted post-implementation focus groups with a randomly selected sub-sample of participants who participated in the intervention and completed their final 6-month appointment in each implementation cycle.

Implementation of the WHC in usual care settings has the potential to reach more vulnerable women and could have a high public health impact if implementation is shown to be effective and sustainable in these real-world settings.

ELIGIBILITY:
Clinic Inclusion Criteria:

* HIV/antenatal clinic or substance abuse treatment clinic
* Located in townships surrounding Cape Town
* Willing to take part in study

Patient Inclusion Criteria:

* Female;
* 18 to 45 years of age;
* Reports use of at least one drug, including alcohol, at least weekly during the previous 3 months;
* Reports unprotected sex with a male partner in the past 6 months;
* Has a positive HIV test result from either the participating health clinic or rehab clinic, or a clinic issued ARV card or ARV medication as proof of positive status;
* Reports the intention to remain in the area for at least the next 6 months;
* Provides informed consent to participate.

Patient Exclusion Criteria:

* Not HIV Positive
* Not willing to do alcohol and drug screening

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 564 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-12-04 (Actual); Study Completion 2018-12-04 (Actual)

PRIMARY OUTCOMES:
Implementation and Service Outcomes: Readiness for appropriate change (appropriateness) | Baseline
  Explore perceived appropriateness of implementing the intervention through qualitative focus groups with clinic staff and patients
Implementation and Service Outcomes: Readiness for appropriate change (appropriateness) | 6-months post-enrollment
  Explore perceived appropriateness of implementing the intervention through qualitative focus groups with clinic staff and patients
Implementation and Service Outcomes: Readiness for appropriate change (appropriateness) | Baseline
  Explore perceived appropriateness of implementing the intervention through clinic staff survey
Implementation and Service Outcomes: Acceptability of the Women's Health CoOp (WHC) intervention | Baseline
  Assess perceived acceptability through qualitative focus groups with clinic staff and patients
Implementation and Service Outcomes: Acceptability of the Women's Health CoOp (WHC) intervention | 6-months post-enrollment
  Assess perceived acceptability through qualitative focus groups with clinic staff and patients
Implementation and Service Outcomes: Acceptability of the Women's Health CoOp (WHC) intervention | Baseline
  Assess perceived acceptability through patient interviews
Implementation and Service Outcomes: Acceptability of the Women's Health CoOp (WHC) intervention | 6-months post-enrollment
  Assess perceived acceptability through patient interviews
Implementation and Service Outcomes: Acceptability of the Women's Health CoOp (WHC) intervention | Baseline
  Assess perceived acceptability through clinic staff survey
Implementation and Service Outcome: Adoption of the Women's Health CoOp (WHC) intervention | Baseline
  Assess adoption of the intervention through qualitative focus groups with clinic staff.
Implementation and Service Outcome: Adoption of the WHC intervention | 6-months post-enrollment
  Assess adoption of the intervention through qualitative focus groups with clinic staff.
Implementation and Service Outcome: Cost | Baseline
  Assess start up and ongoing implementation costs
Implementation and Service Outcome: Cost | 6-months post-enrollment
  Assess start up and ongoing implementation costs
Implementation and Service Outcome: Feasibility | Throughout the period of the study, up to a maximum of one year
  Exposure as measured by the ratio of the number of intervention workshops delivered to participants (a total of two across the intervention window) (compared to the total expected intervention visits. Acceptable retention measured at ≥85% of patients who complete both workshops within the intervention window.
Implementation and Service Outcome: Fidelity | Throughout the study at bimonthly intervals for up to one year
  Observation: fidelity item scores where a 90% or above fidelity rating will indicate acceptable fidelity
Implementation and Service Outcomes: Sustainability | Throughout the period of the study, up to a maximum of one year
  Examine sustainability through qualitative focus groups with clinic staff
Implementation and Service Outcomes: Sustainability | 6 months post-intervention
  Examine sustainability with clinic staff using an adapted TCU Workshop Assessment Follow-up Scale

SECONDARY OUTCOMES:
Antiretroviral Therapy (ART) Initiation and Adherence | Baseline
  Number of participants that received clinical staging, were prescribed and initiated on antiretroviral therapy (ART) and were adhering to ART.
Antiretroviral Therapy (ART) Initiation and Adherence | 6 months post-enrollment
  Number of participants that received clinical staging, were prescribed and initiated on antiretroviral therapy (ART) and were adhering to ART.
Alcohol Use - self-reported frequency and amount | Baseline
  Participants' self-reported frequency and amount of alcohol use will be used to assess recent alcohol use.
Alcohol Use - self-reported frequency and amount | 6 months post-enrollment
  Participants' self-reported frequency and amount of alcohol use will be used to assess recent alcohol use.
Alcohol Use | Baseline
  Breathalyzer test results will be used to assess recent alcohol use.
Alcohol Use | 6 months post-enrollment
  Breathalyzer test results will be used to assess recent alcohol use.
Substance Use | Baseline
  Participants' frequency of benzodiazepines, cocaine, methamphetamine, MDMA, marijuana, and/or mandrax use will be used to assess recent substance use.
Substance Use | 6-months post-enrollment
  Participants' frequency of benzodiazepines, cocaine, methamphetamine, MDMA, marijuana, and/or mandrax use will be used to assess recent substance use.
Substance use | Baseline
  Urine drug screen test results will be used to assess recent use of drugs (benzodiazepines, cocaine, methamphetamine, MDMA, marijuana, and/or mandrax).
Substance use | 6-months post-enrollment
  Urine drug screen test results will be used to assess recent use of drugs (benzodiazepines, cocaine, methamphetamine, MDMA, marijuana, and/or mandrax).
Sexual Risk | Baseline
  Participants' self-reported frequency of condom use.
Sexual Risk | 6-months post-enrollment
  Participants' self-reported frequency of condom use.
Sexual Risk | Baseline
  Participants' self-reported number of sex partners.
Sexual Risk | 6-months post-enrollment
  Participants' self-reported number of sex partners.
Violence/Victimization | Baseline
  Percentages of participants who report being beaten, attacked with a weapon, or forced to have sex.
Violence/Victimization | 6-months post-enrollment
  Percentages of participants who report being beaten, attacked with a weapon, or forced to have sex.
Sexual Communication | Baseline
  The extent to which women have the skills to discuss sexual topics with their partners
Sexual Communication | 6-months post-enrollment
  The extent to which women have the skills to discuss sexual topics with their partners
Relationship Power | Baseline
  The extent to which women and their partners can equitably make decisions together as measured by the Relationship Power Scale (RPS)
Relationship Power | 6-months post-enrollment
  The extent to which women and their partners can equitably make decisions together as measured by the Relationship Power Scale (RPS)

CONTACTS AND LOCATIONS:
Overall Officials: Felicia Browne, ScD, Principal Investigator — RTI International
Locations (2):
- RTI International, Research Triangle Park, North Carolina, United States
- Kheth'Impilo, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Wechsberg WM, Ndirangu JW, Speizer IS, Zule WA, Gumula W, Peasant C, Browne FA, Dunlap L. An implementation science protocol of the Women's Health CoOp in healthcare settings in Cape Town, South Africa: A stepped-wedge design. BMC Womens Health. 2017 Sep 18;17(1):85. doi: 10.1186/s12905-017-0433-8. PMID 28923034
- [Background] Howard BN, Van Dorn R, Myers BJ, Zule WA, Browne FA, Carney T, Wechsberg WM. Barriers and facilitators to implementing an evidence-based woman-focused intervention in South African health services. BMC Health Serv Res. 2017 Nov 21;17(1):746. doi: 10.1186/s12913-017-2669-2. PMID 29157230
- [Result] Wechsberg WM, Browne FA, Ndirangu J, Bonner CP, Kline TL, Gichane M, Zule WA. Outcomes of Implementing in the Real World the Women's Health CoOp Intervention in Cape Town, South Africa. AIDS Behav. 2021 Dec;25(Suppl 3):276-289. doi: 10.1007/s10461-021-03251-7. Epub 2021 Apr 23. PMID 33891233
- [Result] Gichane MW, Wechsberg WM, Ndirangu J, Browne FA, Bonner CP, Grimwood A, Shaikh N, Howard B, Zule WA. Implementation science outcomes of a gender-focused HIV and alcohol risk-reduction intervention in usual-care settings in South Africa. Drug Alcohol Depend. 2020 Oct 1;215:108206. doi: 10.1016/j.drugalcdep.2020.108206. Epub 2020 Aug 1. PMID 32771909
- [Result] Browne FA, Gichane MW, Shangase N, Ndirangu J, Bonner CP, Wechsberg WM. Social Determinants of Alcohol and Other Drug Misuse Among Women Living with HIV in Economically Underserved Communities in Cape Town, South Africa: A Cross-Sectional Study. AIDS Behav. 2023 Apr;27(4):1329-1338. doi: 10.1007/s10461-022-03869-1. Epub 2022 Nov 7. PMID 36344731
- [Result] Gichane MW, Wechsberg WM, Ndirangu J, Howard B, Bonner CP, Browne FA, Zule WA. Sustainability of a gender-focused HIV and alcohol risk-reduction intervention in usual care settings in South Africa: a mixed methods analysis. AIDS Care. 2021 Jan-Dec;33(sup1):11-17. doi: 10.1080/09540121.2021.1966694. Epub 2021 Sep 19. PMID 34538158
- [Result] Ndirangu JW, Gichane MW, Browne FA, Bonner CP, Zule WA, Cox EN, Smith KM, Carney T, Wechsberg WM. 'We have goals but [it is difficult]'. Barriers to antiretroviral therapy adherence among women using alcohol and other drugs living with HIV in South Africa. Health Expect. 2022 Apr;25(2):754-763. doi: 10.1111/hex.13422. Epub 2022 Jan 21. PMID 35060260
- [Result] Washio Y, Browne FA, Ndirangu J, Kline TL, Wechsberg WM. Antiretroviral Therapy (ART) Adherence and Prenatal Alcohol Use among Women Who Are Pregnant with HIV in South Africa. Int J Environ Res Public Health. 2021 Jul 13;18(14):7446. doi: 10.3390/ijerph18147446. PMID 34299897
- [Result] Wechsberg WM, Browne FA, Bonner CP, Washio Y, Howard BN, van der Drift I. Current Interventions for People Living with HIV Who Use Alcohol: Why Gender Matters. Curr HIV/AIDS Rep. 2021 Aug;18(4):351-364. doi: 10.1007/s11904-021-00558-x. Epub 2021 Jun 10. PMID 34110591